CLINICAL TRIAL: NCT02050815
Title: A Phase I, Multicenter, Open-label, Single-dose Study to Assess the Pharmacokinetics of MEK162 in Subjects With Mild, Moderate and Severe Hepatic Impairment
Brief Title: MEK162 in Healthy Subjects With Normal Hepatic Function and Subjects With Impaired Hepatic Function
Acronym: MEK162
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor is terminating the study because the primary objective was achieved after 5 of the 6 subjects were assessed in the final cohort.
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162A2104
Record Dates: First submitted 2014-01-16; First posted 2014-01-31 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Hepatic Impairment
Keywords: MEK162; Hepatic impairment; Healthy subjects
MeSH Terms: interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MEK162 (Experimental): A minimum of 24 subjects (6 subjects per group) will be enrolled. Enrollment into Group 1 (control group with normal hepatic function) should be similar to the enrollment into Group 2, 3 and 4 with respect to age, gender, and body weight. Enrollment into Group 1 will remain open until the enrollment into the mild, moderate, and severe impairment groups are complete with matching controls for comparison. Serum level of total bilirubin and AST will be used to determine which group the hepatic impaired patient will be allocated l. Dosing of the different treatment groups will be staggered. Initially, 6 subjects in Group 1 (normal hepatic function) and 6 subjects in Group 2 will receive a single oral dose of MEK162 on Day 1.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162

SUMMARY:
This study is a phase I, multi-center, open-label, single oral dose, parallel group study to assess the PK and safety of MEK162 in subjects with impaired hepatic function and healthy subjects with normal hepatic function. Subjects will be assigned by hepatic function defined by elevation of serum total bilirubin and serum AST as determined at the screening and baseline visits. The study population will be healthy male and postmenopausal or sterile female subjects who meet all of the inclusion and none of the exclusion criteria. A minimum of 24 evaluable subjects (6 subjects per group) will be enrolled. The groups are: Group 1-healthy volunteers, Group 2-Mild hepatic impairment, Group 3-Moderate hepatic impairment and Group 4-Severe hepatic impairment. Once approved for enrollment, participants will be confined to the facility for 5 days, given a single dose of MEK162 and monitored for safety assessments, labs and PK will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any screening procedures
* Male or female (postmenopausal or sterilized)
* Subject body weight at least 45 kg and a body mass index (BMI) in the range of 18 to 35.0 kg/m2
* Subjects with normal hepatic function must have total bilirubin ≤ upper limit of normal (≤ ULN), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT) and alkaline phosphatase (AP) ≤ ULN, serum creatinine ≤ ULN, serum amylase and lipase ≤ ULN

Additional inclusion criteria for subjects with abnormal liver function determined by elevation of serum total bilirubin are:

* Absolute neutrophil count (ANC) > 1000 cell/mm3
* Hb > 9 mg/dl,
* Platelet count > 30,000/mm3
* Serum creatinine ≤ 1.8 mg/dl
* Otherwise considered healthy and free of significant medical disorders unrelated to the subject's hepatic disorder

Exclusion Criteria:

* Women of child-bearing potential
* Pregnant or nursing (lactating) women
* Subjects with impaired cardiovascular function or clinically significant cardiovascular diseases
* Uncontrolled arterial hypertension despite medical treatment
* History or current evidence of retinal vein occlusion (RVO) or current risk factors of RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes),
* History of Gilbert's syndrome
* Immuno-compromised subjects (including known history/seropositivity of HIV)
* Any surgical or medical condition (other than hepatic impairment) or receiving any pharmacological treatment which might significantly alter the absorption or metabolism of drugs or which may jeopardize the subject in case of participation in the study
* Antecedent of malignancy with the following exceptions: adequately treated basal cell or squamous cell carcinoma of the skin
* Subjects who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Subjects who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure
* History of clinically significant drug allergy
* Prior therapy with a MEK-inhibitor
* Use of an investigational drug within 30 days of screening
* Current smoker or has used tobacco products or products containing nicotine within 7 days prior to dosing of study drug
* Consumption of alcohol within 3 days prior to dosing or during the study

Additional exclusion criteria for subjects with normal hepatic function:

- Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as ALT, AST, GGT, alkaline phosphatase, or serum bilirubin. ALT and AST beyond the normal range before inclusion Presence of impaired renal function as indicated by abnormal creatinine (creatinine clearance < 80 mL/min) values and/or serum creatinine ≥1.8 mg/dL- A positive Hepatitis B or Hepatitis C test result

Additional exclusion criteria for subjects with elevation of serum bilirubin > UNL:

* Symptoms or history of encephalopathy (Grade II or worse) within 4 weeks of study entry
* Clinical evidence of severe ascites requiring intervention
* International normalized ratio (INR) >2.5
* Any evidence of progressive liver disease within the last 3 weeks prior to the screening visit) as indicated by worsening of clinical manifestations (i.e.: ascites, encephalopathy) and/or laboratories abnormalities (liver transaminases, alkaline phosphatase and GGT or a ≥ 50% worsening of serum bilirubin or prothrombin time)
* History of surgical portosystemic shunt with complications (i.e. hepatic encephalopathy, heart failure)
* Active bleeding during the last 28 days prior to dosing including variceal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
PK parameters assessed by Tmax | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120
  Blood pharmacokinetic samples will be collects at various timepoints to assess the MEK162 concentration levels. MEK162 concentrations and preliminary PK parameters will be analyzed in the two groups to determine if a dose adjustment is required in patients with moderate hepatic impairment
PK parameters assessed by Cmax | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120
  Blood pharmacokinetic samples will be collects at various timepoints to assess the MEK162 concentration levels. MEK162 concentrations and preliminary PK parameters will be analyzed in the two groups to determine if a dose adjustment is required in patients with moderate hepatic impairment
PK parameters assessed by AUCinf | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120
  Blood pharmacokinetic samples will be collects at various timepoints to assess the MEK162 concentration levels. MEK162 concentrations and preliminary PK parameters will be analyzed in the two groups to determine if a dose adjustment is required in patients with moderate hepatic impairment
PK parameters assessed by AUC0last | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120
  Blood pharmacokinetic samples will be collects at various timepoints to assess the MEK162 concentration levels. MEK162 concentrations and preliminary PK parameters will be analyzed in the two groups to determine if a dose adjustment is required in patients with moderate hepatic impairment

SECONDARY OUTCOMES:
Relationship between PK parameters versus hepatic function laboratory parameters | Screening, Baseline, Day 2, Day 6 (Day of discharge)
  To explore the relationship between hepatic liver function and PK. Pharmacokinetic parameters will be correlated to hepatic lab parameters.
Number of subjects with adverse events as a measure of safety and tolerability | Screening, Baseline, Day 2, Day 6 (Day of discharge)
  Adverse events based on the Common Terminology Criteria for Adverse Events (CTCAE) grade (severity) and frequency, and other safety data

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - DaVita Clinical Research-Denver, Lakewood, Colorado
  - Clinical Pharmacology of Miami (CPMI), Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Kansas City Research Institute, LLC, Kansas City, Missouri

REFERENCES:
- [Derived] Piscitelli J, Hahn E, Wollenberg L, Chavira R, Del Frari L, Reddy MB. Pharmacokinetics of Binimetinib in Participants with Hepatic Impairment. Clin Pharmacokinet. 2025 Aug;64(8):1217-1230. doi: 10.1007/s40262-025-01509-0. Epub 2025 Jun 23. PMID 40549341